CLINICAL TRIAL: NCT04253925
Title: Effect of Global Postural Correction Exercises on Stress Urinary Incontinence During Pregnancy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, lecture of biomechanics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/00976
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Stress Urinary Incontinence
Keywords: Kegel exercise; Postural Correction; Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- global postural correction exercises (Experimental): global postural correction exercises in addition to Kegel exercises
  Interventions: Other: Kegel exercises
- Kegel exercises (Active Comparator): only Kegel exercises
  Interventions: Other: Kegel exercises

INTERVENTIONS:
Other: Kegel exercises — global postural correction exercises

SUMMARY:
Background: One of the many consequences of pregnancy that may negatively affect a woman's quality of life is stress urinary incontinence caused by activities of daily living especially those associated with increased intraabdominal pressure. Objective: This study aimed to investigate the effect of global postural correction exercises on stress urinary incontinence among pregnant women. Participants and Methods: Forty primigravida women (aged between 30-39 years), with a single fetus, diagnosed with stress urinary incontinence participated in the study. Participants were assigned randomly into two groups: Study group (group A; n=20) and control group (group B; n=20). The participants were tested twice, before and after a 12-week period, during which group A received global postural correction exercises in addition to Kegel exercises, while group B performed only Kegel exercises. A perineometer was used to evaluate the change in vaginal squeeze pressure both before and after conducting the study. Urogenital Distress Inventory Questionnaire (UDI-6) was used to assess changes in incontinence severity symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Forty primigravida women with singleton fetus in their third trimester and diagnosed with pregnancy related SUI participated in this study.

All participants suffered from a mild to moderate grade of SUI identified by clinical grading (Ingelman-Sundberg) (Wlazlak et al., 2015) as follows: Grade I (mild), the leakage of urine occurs on straining; and grade II (moderate), the leakage occurs following abrupt movement

Exclusion Criteria:

* Females were excluded from the study if they had severe grade SUI; infections in their lower urinary tract; neurological conditions; gestational diabetes; and chronic chest diseases. Females who smoked, used any medications or medical/surgical interventions for SUI, or who suffered any other type of urinary incontinence were also excluded from the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
strength of pelvic floor muscle | change from Baseline strength of pelvic floor muscle at 12-weeks

SECONDARY OUTCOMES:
Urogenital Distress Inventory Questionnaire | change from Baseline Urogenital Distress Inventory Questionnaire (UDI-6) at 12-weeks

IPD SHARING:
Plan to Share IPD: Undecided